CLINICAL TRIAL: NCT02211170
Title: The Effect of Single Oral Dose BIRB 796 BS (50 and 600 mg) on Endotoxin-induced Inflammatory Responses in Healthy Human Subjects. A Placebo-controlled, Randomised, Parallel, Double-blinded Study.
Brief Title: Effect of Single Oral Dose BIRB 796 BS on Endotoxin-induced Inflammatory Responses in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.4
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Lipopolysaccharides

ARMS (3):
- BIBR 796 BS, low dose (Experimental)
  Interventions: Drug: BIBR 796 BS, low dose; Drug: Lipopolysaccharide
- BIBR 796 BS, high dose (Experimental)
  Interventions: Drug: BIBR 796 BS, high dose; Drug: Lipopolysaccharide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Lipopolysaccharide

INTERVENTIONS:
Drug: BIBR 796 BS, low dose
  Arms: BIBR 796 BS, low dose
Drug: BIBR 796 BS, high dose
  Arms: BIBR 796 BS, high dose
Drug: Placebo
  Arms: Placebo
Drug: Lipopolysaccharide — Lipopolysaccharide (LPS) for endotoxin challenge

SUMMARY:
Study to determine the effect of a single dose BIRB 796 BS on systemic inflammatory responses induced by endotoxin in healthy humans

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice and local legislation
* Age ≥18 and ≤ 35 years
* Broca ≥- 20 % and ≤ + 20%
* Able to communicate well with the investigator and to comply with study requirements

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and EKG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections within 14 days of enrolment
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 3 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 ml (< 2 month prior to administration or during the trial)
* Excessive physical activities (< 24 hours prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* History of any familial bleeding disorder
* Weight > 150 kg
* Prior confirmed or suspected receipt of a monoclonal antibody

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-02; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Reduction of tumour necrosis factor alpha (TNFα) concentration | up to 2 days

SECONDARY OUTCOMES:
Reduction of pro-inflammatory cytokines (IL-6, IL-8, G-CSF) | up to 2 days
Reduction of anti-inflammatory cytokine and cytokine inhibitors (IL-10, IL-12p40, soluble TNF receptor (sTNFr) type 1, IL-1ra) | up to 2 days
Reduction of Acute Phase Proteins (C-reactive protein, Haptoglobin) | up to 2 days
Reduction of Endothelial Activation Markers (von Willebrand Factor, soluble E-selectin) | up to 2 days
Reduction of Granulocyte Responses (white blood cell (WBC) count with differential, elastase, elastase-á1-antitrypsin complexes) | up to 2 days
Reduction of flow Cytometry Cell Surface Markers (Mac-1 (macrophage-1 antigen), L-Selectin) | up to 2 days
Reduction of ex vivo p38 mitogen-activated protein kinase (MAPK) phosphorylation activity | up to 2 days
Occurence and severity of with chills, nausea, vomiting, abdominal pain, backache, headache, myalgia, fever | up to 2 days
Number of patients with clinically significant changes in vital signs (pulse rate, systolic and diastolic blood pressure, temperature) | up to 14 days
Number of patients with abnormal changes in laboratory parameters | up to 14 days
Number of patients with adverse events | up to 14 days
Assessment of Global Clinical Tolerability on a 4-point scale | after 14 days
Maximum plasma concentration (Cmax) | up to 27 hours after drug administration
Time at which Cmax occurred (tmax) | up to 27 hours after drug administration
Elimination half life (t1/2), | up to 27 hours after drug administration
Area under the plasma concentration-time curve for different time points(AUC) | up to 27 hours after drug administration
Apparent clearance (CL/F) | up to 27 hours after drug administration
Elimination rate constant (λz) | up to 27 hours after drug administration
Mean residence time (MRT) | up to 27 hours after drug administration
Apparent volume of distribution (Vz/F) | up to 27 hours after drug administration